CLINICAL TRIAL: NCT06340217
Title: The Efficacy and Safety of WMT in the Treatment of Diabetic Gastroparesis: A Multicenter, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Washed Microbiota Transplantation for Diabetic Gastroparesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WMT-GDP-RCT
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Gastroparesis
Keywords: washed microbiota transplantation; diabetic gastroparesis; randomized controlled trial; transendoscopic enteral tube; microbiota medicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The patient will receive WMT once daily for a duration of 2 days
  Interventions: Other: washed microbiota transplantation
- Control (Placebo Comparator): The patient will receive a placebo of equal volume once daily for a duration of 2 days
  Interventions: Other: placebo

INTERVENTIONS:
Other: washed microbiota transplantation — Washed microbiota transplantation refers to the infusion of washed microbiota from healthy donor into patients' gastrointestinal tract. Participants will receive two doses of WMT for DGP.
  Arms: Treatment
Other: placebo — A carrier fluid with matching volume and consistent appearance to the infusion of washed microbiota.
  Arms: Control

SUMMARY:
This is a randomized controlled trial to explore the efficacy and safety of washed microbiota transplantation (WMT) for diabetic gastroparesis (DGP) patients.

DETAILED DESCRIPTION:
At least 44 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. Data of demographic characteristics, Gastroparesis Cardinal Symptom Index (GCSI), Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM), Gastroparesis Core Symptom Daily Diary (GCS-DD), Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QoL), and clinical outcomes will be collected. After treatment, they will enter the follow-up period for efficacy and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to enter the study:

1. Diagnosed with diabetes for over 1 year;
2. Accompanied by symptoms such as abdominal bloating, early satiety, persisting for at least 3 months, with a GCSI Total Score greater than/equal to 2.3;
3. Objective evidence of delayed gastric emptying within the past 3 months, including but not limited to scintigraphic gastric emptying or gastric ultrasound;
4. Upper gastrointestinal obstructive lesions were ruled out by imaging or endoscopic examination within the past 3 months;
5. Males and nonpregnant, non-breastfeeding females who are aged more than 18 years and sign the informed consent form;
6. The subject or his/her legal representative gives informed consent, fully understands the purpose of the study, is able to communicate effectively with the investigator, and comprehends and complies with the requirements set forth in the study.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria must be excluded from the study:

Subjects who:

1. Have any upper gastrointestinal pathology other than diabetic gastroparesis that would require therapy other than that provided in this trial;
2. Have a prior history of gastric surgery, including but not limited to gastric bypass, gastrectomy, gastric banding, pyloroplasty, fundoplication, or vagotomy in past 1 year;
3. Have any organic/neurological disease that is suspected to be causing gastroparesis, other than diabetes;
4. Have been using medications affecting gastrointestinal motility, such as GLP-1 agonists;
5. Have contraindications for intestinal tubing;
6. Have a history of medication that regulate intestinal microbiome in last 48 hours;
7. Have serious diabetic complications need immediately be dealt, such as diabetic ketoacidosis
8. Have poor lung function and those deemed by the investigator to be affected by the study treatment, such as during COPD exacerbations;
9. Have any of the following abnormalities in cardiac function and cardiac performance:

   * Cardiac function rating≥Ⅲ according to New York Heart Association (NYHA);
   * New myocardial infarction or unstable angina pectoris within 6 months;
   * Electrocardiogram indicated prolonged QTc interval (male QTc≥450ms, female QTc≥470ms);
   * requiring drug intervention (more than Ⅱ atrioventricular block).
10. Have preexisting hepatic disease that meets Child-Pugh Class B (moderate; total score 7 to 9 points) or C (severe; total score 10 to 15 points);
11. Kidney disease with KDIGO stage 3b (GFR<45 ml/min/1.73m2) or above;
12. Have infectious diseases such as active hepatitis (requiring long-term use of drugs), HIV or active tuberculosis;
13. Have a history of drug abuse, alcoholism (defined as consuming more than 14 units per week, with 1 unit equivalent to 360 mL of beer, 45 mL of 40% alcohol, or 150 mL of wine), or substance misuse;
14. Other significant systemic illnesses, such as malignant tumors;
15. Have other situations in which the investigator deems it inappropriate to participate in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of DGP with symptom relief after the procedure. | Four-week post-WMT
  Detailed evaluation content of efficacy rate of symptom: Symptom relief is defined as a decrease of at least 50% in the total Gastroparesis Cardinal Symptom Index (GCSI).

SECONDARY OUTCOMES:
The extent of change observed in GCSI of participants; | One-week, Two-week and Eight-week post-WMT
  The GCSI consists of nine items and three subscales to measure symptoms related to gastroparesis. The nausea/vomiting subscale consists of the following three items: nausea, retching, and vomiting. The postprandial fullness/early satiety subscale consists of the following four items: stomach fullness, inability to finish a normal-sized meal, feeling excessively full after meals, and loss of appetite.
The extent of change observed in Gastroparesis Core Symptom Daily Diary (GCS-DD) of participants; | One-week, Two-week, Four-week and Eight-week post-WMT
  GCS-DD consists of 13 items for evaluating the core symptom for past 24 hours.
The extent of change observed in Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM) of participants; | One-week, Two-week, Four-week and Eight-week post-WMT
  Questionnaire was developed to measure specific symptoms of patients with upper gastrointestinal disorders. It records 20 symptoms (6 subscales) and assesses their severity within the 2 weeks prior to the test. Subscale scores are calculated by averaging across items comprising the subscale; scores vary from 0 (none or absent) to 5 (very severe). The PAGI-SYM subscale scores have good internal consistency and test-retest reliability.
The extent of change observed in Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QoL) of participants; | One-week, Two-week, Four-week and Eight-week post-WMT
  The PAGI-QoL contains 30 items with five subscales:
  (1) daily activities (1-10); (2) clothing (11-12); (3) diet/food habits (13-19); (4) relationship (20-22); (5) psychological well-being and distress (23-30). Subscale scores are calculated by averaging the item responses.
The extent of change observed in electrogastrogram (EGG) of participants; | One-week, Two-week, Four-week and Eight-week post-WMT
  The frequency of gastric electric waves will be evaluated by EGG.
The extent of change observed in electrogastrogram (EGG) of participants; | One-week, Two-week, Four-week and Eight-week post-WMT
  The amplitude of gastric electric waves will be evaluated by EGG.
The extent of change observed in gastrointestinal ultrasound (GIUS) of participants; | One-week, Two-week, Four-week and Eight-week post-WMT
  The half gastric emptying time will be evaluated by GIUS.
The incidence rate of adverse events; | One-week, Two-week, Four-week and Eight-week post-WMT
  The number of adverse reactions reported by subjects in the WMT group from the start of treatment to the end of follow-up, divided by the total number of WMT treatments.
The changes in gut microbiota composition and metabolites before and after treatment. | One-week, Two-week, Four-week and Eight-week post-WMT
  The 16s-RNA or meta-analysis of gut microbiota will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shin AS, Camilleri M. Diagnostic assessment of diabetic gastroparesis. Diabetes. 2013 Aug;62(8):2667-73. doi: 10.2337/db12-1706. No abstract available. PMID 23881199
- [Background] Ye Y, Jiang B, Manne S, Moses PL, Almansa C, Bennett D, Dolin P, Ford AC. Epidemiology and outcomes of gastroparesis, as documented in general practice records, in the United Kingdom. Gut. 2021 Apr;70(4):644-653. doi: 10.1136/gutjnl-2020-321277. Epub 2020 Jun 3. PMID 32493829
- [Background] Aswath GS, Foris LA, Ashwath AK, Patel K. Diabetic Gastroparesis. 2023 Mar 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK430794/ PMID 28613545
- [Background] Liu J, Liu M, Chai Z, Li C, Wang Y, Shen M, Zhuang G, Zhang L. Projected rapid growth in diabetes disease burden and economic burden in China: a spatio-temporal study from 2020 to 2030. Lancet Reg Health West Pac. 2023 Feb 3;33:100700. doi: 10.1016/j.lanwpc.2023.100700. eCollection 2023 Apr. PMID 36817869
- [Background] Camilleri M, Kuo B, Nguyen L, Vaughn VM, Petrey J, Greer K, Yadlapati R, Abell TL. ACG Clinical Guideline: Gastroparesis. Am J Gastroenterol. 2022 Aug 1;117(8):1197-1220. doi: 10.14309/ajg.0000000000001874. Epub 2022 Jun 3. PMID 35926490
- [Background] Vosoughi K, Ichkhanian Y, Benias P, Miller L, Aadam AA, Triggs JR, Law R, Hasler W, Bowers N, Chaves D, Ponte-Neto AM, Draganov P, Yang D, El Halabi M, Sanaei O, Brewer Gutierrez OI, Bulat RS, Pandolfino J, Khashab M. Gastric per-oral endoscopic myotomy (G-POEM) for refractory gastroparesis: results from an international prospective trial. Gut. 2022 Jan;71(1):25-33. doi: 10.1136/gutjnl-2020-322756. Epub 2021 Mar 19. PMID 33741641
- [Background] Ragi O, Jacques J, Branche J, Leblanc S, Vanbiervliet G, Legros R, Pioche M, Rivory J, Chaussade S, Barret M, Wallenhorst T, Barthet M, Kerever S, Gonzalez JM. One-year results of gastric peroral endoscopic myotomy for refractory gastroparesis: a French multicenter study. Endoscopy. 2021 May;53(5):480-490. doi: 10.1055/a-1205-5686. Epub 2020 Jul 21. PMID 32575130
- [Background] Martinek J, Hustak R, Mares J, Vackova Z, Spicak J, Kieslichova E, Buncova M, Pohl D, Amin S, Tack J. Endoscopic pyloromyotomy for the treatment of severe and refractory gastroparesis: a pilot, randomised, sham-controlled trial. Gut. 2022 Nov;71(11):2170-2178. doi: 10.1136/gutjnl-2022-326904. Epub 2022 Apr 25. PMID 35470243
- [Background] Abdelfatah MM, Noll A, Kapil N, Shah R, Li L, Nustas R, Li B, Luo H, Chen H, Xia L, Mekaroonkamol P, Shahnavaz N, Keilin S, Willingham F, Christie J, Cai Q. Long-term Outcome of Gastric Per-Oral Endoscopic Pyloromyotomy in Treatment of Gastroparesis. Clin Gastroenterol Hepatol. 2021 Apr;19(4):816-824. doi: 10.1016/j.cgh.2020.05.039. Epub 2020 May 22. PMID 32450364
- [Background] Wang Y, Zhang S, Borody TJ, Zhang F. Encyclopedia of fecal microbiota transplantation: a review of effectiveness in the treatment of 85 diseases. Chin Med J (Engl). 2022 Aug 20;135(16):1927-1939. doi: 10.1097/CM9.0000000000002339. PMID 36103991
- [Background] Li Y, Liu Q, Zhang L, Zou J, He R, Zhou Y, Qian C, Zhu Y, Chen R, Zhang Y, Cai P, Wang M, Shao W, Ji M, Wu H, Zhang F, Liu Z, Liu Y. Washed microbiota transplantation reduces glycemic variability in unstable diabetes. J Diabetes. 2024 Feb;16(2):e13485. doi: 10.1111/1753-0407.13485. Epub 2023 Oct 17. PMID 37846600
- [Background] Ng SC, Xu Z, Mak JWY, Yang K, Liu Q, Zuo T, Tang W, Lau L, Lui RN, Wong SH, Tse YK, Li AYL, Cheung K, Ching JYL, Wong VWS, Kong APS, Ma RCW, Chow EYK, Wong SKH, Ho ICH, Chan PKS, Chan FKL. Microbiota engraftment after faecal microbiota transplantation in obese subjects with type 2 diabetes: a 24-week, double-blind, randomised controlled trial. Gut. 2022 Apr;71(4):716-723. doi: 10.1136/gutjnl-2020-323617. Epub 2021 Mar 30. PMID 33785557
- [Background] Yang J, Yang X, Wu G, Huang F, Shi X, Wei W, Zhang Y, Zhang H, Cheng L, Yu L, Shang J, Lv Y, Wang X, Zhai R, Li P, Cui B, Fang Y, Deng X, Tang S, Wang L, Yuan Q, Zhao L, Zhang F, Zhang C, Yuan H. Gut microbiota modulate distal symmetric polyneuropathy in patients with diabetes. Cell Metab. 2023 Sep 5;35(9):1548-1562.e7. doi: 10.1016/j.cmet.2023.06.010. Epub 2023 Jul 13. PMID 37451270
- [Background] Camilleri M, Chedid V, Ford AC, Haruma K, Horowitz M, Jones KL, Low PA, Park SY, Parkman HP, Stanghellini V. Gastroparesis. Nat Rev Dis Primers. 2018 Nov 1;4(1):41. doi: 10.1038/s41572-018-0038-z. PMID 30385743
- [Background] Huang Y, Guo Y, Li X, Xiao Y, Wang Z, Song L, Ren Z. Effects of Lactiplantibacillus plantarum GUANKE on Diphenoxylate-Induced Slow Transit Constipation and Gut Microbiota in Mice. Nutrients. 2023 Aug 26;15(17):3741. doi: 10.3390/nu15173741. PMID 37686774
- [Background] Prochazkova N, Falony G, Dragsted LO, Licht TR, Raes J, Roager HM. Advancing human gut microbiota research by considering gut transit time. Gut. 2023 Jan;72(1):180-191. doi: 10.1136/gutjnl-2022-328166. Epub 2022 Sep 28. PMID 36171079
- [Background] Falony G, Joossens M, Vieira-Silva S, Wang J, Darzi Y, Faust K, Kurilshikov A, Bonder MJ, Valles-Colomer M, Vandeputte D, Tito RY, Chaffron S, Rymenans L, Verspecht C, De Sutter L, Lima-Mendez G, D'hoe K, Jonckheere K, Homola D, Garcia R, Tigchelaar EF, Eeckhaudt L, Fu J, Henckaerts L, Zhernakova A, Wijmenga C, Raes J. Population-level analysis of gut microbiome variation. Science. 2016 Apr 29;352(6285):560-4. doi: 10.1126/science.aad3503. Epub 2016 Apr 28. PMID 27126039
- [Background] Asnicar F, Leeming ER, Dimidi E, Mazidi M, Franks PW, Al Khatib H, Valdes AM, Davies R, Bakker E, Francis L, Chan A, Gibson R, Hadjigeorgiou G, Wolf J, Spector TD, Segata N, Berry SE. Blue poo: impact of gut transit time on the gut microbiome using a novel marker. Gut. 2021 Sep;70(9):1665-1674. doi: 10.1136/gutjnl-2020-323877. Epub 2021 Mar 15. PMID 33722860
- [Background] Larraufie P, Martin-Gallausiaux C, Lapaque N, Dore J, Gribble FM, Reimann F, Blottiere HM. SCFAs strongly stimulate PYY production in human enteroendocrine cells. Sci Rep. 2018 Jan 8;8(1):74. doi: 10.1038/s41598-017-18259-0. PMID 29311617
- [Background] Dimidi E, Christodoulides S, Scott SM, Whelan K. Mechanisms of Action of Probiotics and the Gastrointestinal Microbiota on Gut Motility and Constipation. Adv Nutr. 2017 May 15;8(3):484-494. doi: 10.3945/an.116.014407. Print 2017 May. PMID 28507013
- [Background] Horvath VJ, Putz Z, Izbeki F, Korei AE, Gero L, Lengyel C, Kempler P, Varkonyi T. Diabetes-related dysfunction of the small intestine and the colon: focus on motility. Curr Diab Rep. 2015 Nov;15(11):94. doi: 10.1007/s11892-015-0672-8. PMID 26374571